CLINICAL TRIAL: NCT04119141
Title: Benefit of Tin Filter in Regards to Image Quality and Radiation Dose in CT Scan
Brief Title: Benefit of Tin Filter in Regards to Image Quality and Radiation Dose in CT Scan Study of Pulmonary Parenchyma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr Béatrice Daoud (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 2018-A00918-47
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Tin X Ray; Pulmonary Parenchyma
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arm (Active Comparator): the first acquisition will be carried out without a tin filter in supine position and the second with tin filter in procubitus.
  Interventions: Diagnostic Test: X ray imaging
- Tin filter Arm (Experimental): the first acquisition will be carried out with tin filter in supine position and the second without tin filter in procubitus.
  Interventions: Diagnostic Test: X ray imaging

INTERVENTIONS:
Diagnostic Test: X ray imaging — Acquisition:
  * 140 kVp,
  * 1/2 mAs/kg,
  * Pitch: 1.35,
  * Rotation time: 0.5 sec.
  Reconstruction:
  * I70f filter, 3 iteration loops,
  * Cutting thickness 1 mm/0.7 mm
  * Fenestration: C -600/W 1600
  * Field of view (Size, x & y coordinates) identical on both acquisitions.

SUMMARY:
Main objective: to demonstrate that the diagnostic quality associated with the acquisition mode with tin filter, evaluated in a subjective way, is not inferior to that associated with the acquisition mode without filter.

DETAILED DESCRIPTION:
The chest x-ray is the first-line exam for the study of pulmonary parenchyma. Nevertheless, it does not make it possible to reveal all pulmonary pathologies, and in particular those of very small sizes. Thanks to its very high spatial resolution and contrast resolution, the scanner is able to detect all infra-millimetric pathologies of the pulmonary parenchyma but also mediastinal pathologies that could not have been seen on the standard x-ray.

This study fits into the context of pleural pathology screening for patients exposed to asbestos in their professional environment.

Today, the chest CT scan in millimetric sections isth e standardised method used in the context of this screening.Tin filtration is an additional filtration at the output of the X-ray tube made available on premium Siemens scanners. In diagnostic medical imaging, the photon beam has an energetic spectrum ranging from 0 to 150 keV. However the weak energies do not participate in the formation of the image but, on the other hand, to the overall radiation of the patient. The purpose of the addition of the tin filter is to be able to suppress, at the output of the tube, all low and medium energy levels, only allowing high energy levels to pass through. A previous study comparing the same group of patients on two different machines (one with tin filtration, one without tin filtration) showed a significant decrease in the radiation dose; nevertheless, a certain number of parameters differed between the two scanners used. In order to get rid of the different biases encountered on previous published studies, we propose to carry out this study on the same machine, by activating and deactivating tin filtration, all other parameters of acquisition and reconstruction of the image being equal in all respects.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over.
* Patient referred for chest CT scan in the context of screening or monitoring of occupational exposure to asbestos.
* Patient with health insurance or beneficiary of a social security scheme.
* Patient having given their express consent.

Exclusion Criteria:

* Woman who is pregnant or likely to be pregnant.
* Lactating or parturient women
* Minors.
* Protected patients: Adults under trusteeship, guardianship or other legal protection, deprived of liberty by judicial or administrative decision; hospitalised without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Likert score scale score | 1 hour
  Primary endpoint: score obtained on the Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé d'Antony Antony, Antony, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided